CLINICAL TRIAL: NCT00461864
Title: Diagnosis of Occult Hip Fractures With Ultrasound
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Other Study IDs: HIPUS-1
Record Dates: First submitted 2007-04-16; First posted 2007-04-18 (Estimated); Last update posted 2007-04-18 (Estimated); Status verified 2007-03

CONDITIONS: Hip Fractures; Occult Fractures
Keywords: fracture; occult; hip
MeSH Terms: conditions — Hip Fractures; Fractures, Closed; Fractures, Bone

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: ultrasound examination of the hip

SUMMARY:
occult hip fractures present to the emergency room with a history of trauma,a painful hip and normal X-ray. these patients usually undergo other imaging modalities such as CT scans, MRI, or bone scans.

In this study we check the sensitivity and specificity of a directed ultrasound examination of the hip joint in diagnosing or excluding a hip fracture. We also compare the results of ultrasound examination by the orthopedic surgeon in the emergency room versus the consultant radiologist.

The patients undergo bone scans or CT to make the diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* patients over age of 50 with clinical suspicion of a hip fracture

Exclusion Criteria:

* previous fracture or surgical intervention in the hip
* pregnancy
* flexion contracture of hip

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2007-04

CONTACTS AND LOCATIONS:
Overall Officials: Alon Burg, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel